CLINICAL TRIAL: NCT02405468
Title: Identification of the Blood Microbiota in Patient Suffering From Myocardial Infraction
Acronym: FLORINF
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 12 387 02; 2013-A00337-38 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Disease; Myocardial Infarction
Keywords: blood microbiota; coronary disease; myocardial infarction
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case: patients with a myocardial infarction within one month to one year before the inclusion
- control: patients without history of myocardial infarction, free of coronary disease in the view of one of the following test performed within one year before the inclusion : Effort test Echocardiographic stress test Myocardial perfusion scintigraphy Coronarography with >= 2 major cardiovascular risk factors :
  * Treated hypertension
  * Treated dyslipidemia
  * Current smoking
  * Diabetes mellitus

SUMMARY:
The investigators want to compare blood microbiota profile between patients with documented coronary lesions and patients free of coronary disease.

ELIGIBILITY:
Inclusion Criteria:

* Cases : patients who have had a myocardial infarction within one month to one year before the inclusion
* Controls : patients without history of myocardial infarction, free of coronary disease in the view of one of the following tests performed within one year before the inclusion :

Effort test Echocardiographic stress test Myocardial perfusion scintigraphy Coronarography with >= 2 major cardiovascular risk factors:

1. Treated hypertension,
2. Treated dyslipidemia
3. Current smoking
4. Diabetes mellitus

Exclusion Criteria:

* Infectious disease within one week before the inclusion
* Immunocompromised patients
* Antibiotic treatment within one month before the inclusion
* Chronic viral infection
* Chronic inflammatory intestinal bowel disease
* Renal failure (estimated glomerular filtration rate< 50 ml/min//1.73 m2)
* Pregnancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: case : patients who have had a myocardial infarction within one month to one year before the inclusion controls : patients without history of myocardial infarction, free of coronary disease in the view of one of the following tests performed within one year before the inclusion Effort test Echocardiographic stress test Myocardial perfusion scintigraphy Coronarography with >= 2 major cardiovascular risk factors:
  * Treated hypertension,
  * Treated dyslipidemia
  * Current smoking
  * Diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
blood bacterial 16s rDNA bacterial gene concentration | 12 months
  compare blood bacterial 16s rDNA bacterial gene concentration

SECONDARY OUTCOMES:
blood microbiota profile | 12 months
  compare blood microbiota profile as assessed at all taxonomic levels of interest (genus, family, order, class, phylum)

OTHER OUTCOMES:
lipid profile | 12 months
  Obtain an accurate lipid profile with a new technic of microelectrophoresis(Lipoprint)
functional HDL | 12 months
  Analyse the functional qualities of the HDL from the serum
microARN profile | 12 months
  Search a microARN profile corresponding to the coronary heart disease
Serum Bank and DNA Bank | 10 years
  Form a Serum Bank and a DNA Bank for potential future analysis guided by microARN research
modifications of the blood microbiota | 12 months
  Analyse modification of the blood microbiota in the case and the control

CONTACTS AND LOCATIONS:
Overall Officials: Meyer Elbaz, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amar J, Lelouvier B, Servant F, Lluch J, Burcelin R, Bongard V, Elbaz M. Blood Microbiota Modification After Myocardial Infarction Depends Upon Low-Density Lipoprotein Cholesterol Levels. J Am Heart Assoc. 2019 Oct;8(19):e011797. doi: 10.1161/JAHA.118.011797. Epub 2019 Sep 28. PMID 31566105